CLINICAL TRIAL: NCT05526573
Title: Diagnostic Yeld of Ultrathin Bronchoscopy in Peripheral Pulmonary Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Alberto Fantin, Principal Investigator, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: 4393
Record Dates: First submitted 2022-08-28; First posted 2022-09-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Lung Cancer; Lung; Node; Lung Diseases; Lung TB; Lung Adenocarcinoma; Lung Transplant Rejection
Keywords: NSCLC; Lung nodule
MeSH Terms: conditions — Lung Neoplasms; Lung Diseases; Tuberculosis, Pulmonary; Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrathin bronchoscopy (MP190F; Olympus Medical Systems, Tokyo, Japan) — Fluoroscopy + RP-EBUS and consecutive lesion sampling by TBNA and/or TBB

SUMMARY:
The use of an ultrathin bronchoscope (UB) has recently been introduced in the diagnosis of peripheral lung lesions. The use of the UB can be supported by navigation systems such as fluoroscopy, ultrasound guidance, electromagnetic navigation, or other technologies, which have complementary potential. Further navigation techniques are still under study. The use of ultrathin instrumentation has already been shown to significantly reduce procedural times compared to traditional instrumentation.

The purpose of the study is to prospectively evaluate the institutional experience of different third-level hospital centers with the use of a UB (MP190F; Olympus Medical Systems, Tokyo, Japan) for sampling peripheral lung lesions by means of transbronchial needle aspiration (TBNA) or transbronchial biopsy (TBB), performed after fluoroscopic navigation and simultaneous radial probe-endobronchial ultrasound (RP-EBUS) assessment.

Design: multicentric, observational study.

ELIGIBILITY:
Inclusion criteria:

* Candidate for a diagnostic procedure for a new peripheral lung lesion or re-biopsy;
* Tissue sampling of the peripheral lesion performed only with UB;
* The patient's ability to understand the individual characteristics and consequences of the clinical study;
* Males and females of any ethnicity;
* Subjects who have given their informed consent to use their clinical data for research purposes.

Exclusion criteria:

* Inability to give informed consent or understand its contents;
* Unavailability of tomographic imaging;
* Failure to use RP-EBUS or fluoroscopic guidance during the procedure;
* Failure to use R.O.S.E. by the pulmonologist or pathologist during the procedure;
* Tissue sampling on the same peripheral lesion using an instrument of a different caliber in replacement or in association;
* Any other significant illness or disorder that, in the investigator's opinion, may put the patient at risk due to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential screening aimed at recruitment. Enrollment of patients undergoing diagnostic bronchoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the overall diagnostic accuracy | Within 12 months from the procedure
  Sensitivity, specificity, positive predictive value, negative predictive value

SECONDARY OUTCOMES:
Agreement between the definitive pathological result and the rapid on-site evaluation (R.O.S.E.) | Within 15 days from the procedure
  Comparison (% of concordant and % of discordant results) between R.O.S.E. (performed during the procedure by the pulmonologist or by the pathologist) and the final result obtained after the evaluation (by the pathologist) of the samples taken.
Evaluation of patient satisfaction at the end of the procedure (Likert scale in relation to the memory of the procedure and the willingness to repeat it in the future.) | Same day of the procedure
  Patients will undergo two satisfaction questionnaires, set according to Likert scale, at the end of the endoscopic procedure.
Correlation between the type of anesthesia, the characteristics of the lesion, the procedural dynamics and diagnostic accuracy | Within 12 months from the procedure
Correlation between the type of anesthesia, the characteristics of the lesion, the procedural dynamics and patient satisfaction | Same day of the procedure
  Correlations will be made between the anesthetic, radiological and procedural parameters with respect to the answers obtained in the satisfaction questionnaires.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Pneumologia, Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - Pneumologia, Arcispedale S. Maria Nuova, Reggio Emilia
  - Pneumologia, ASUFC, Az. Osp. Santa Maria della Misericordia, Udine